CLINICAL TRIAL: NCT04262583
Title: Assessment of adherenCe tO Medical theraРy and Its infLuence on Long-term Outcomes In pAtieNts With Chronic Heart failurE in the Outpatient Registry
Brief Title: Assessment of adherenCe tO Medical theraРy and Its infLuence on Long-term Outcomes In pAtieNts With Heart Failure
Acronym: COMPLIANCE
Status: Completed | Type: Observational
Sponsor: National Research Center for Preventive Medicine (Other Government)
Responsible Party: Sponsor
Organization: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Other Study IDs: 09062019
Record Dates: First submitted 2020-02-07; First posted 2020-02-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure, adherence, registry
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this prospective cohort study is to assess the adherenсe to medical therapy and its influence on long-term outcomes in patients with chronic heart failure in the outpatient registry

DETAILED DESCRIPTION:
Registry PROFILE is a patients database with cardiovascular diseases who consistently apply to the specialized cardiology department of the "National Medical Research Center for Preventive Medicine" for consultation or to assess their possible participation in clinical trials The purpose of this study is to assess adherence to medical therapy and its impact on long-term outcomes in patients with chronic heart failure enrolled to PROFILE registry from 01 January 2016 to 01 July 2020. The patients who were enrolled between 01 January 2016 to 01 December 2019 will be invited to clinical visit by phone. For patients who will join PROFILE registry after 01 December 2019 the first visit of this study is the day of enrollment to PROFILE registry.

The first visit (V1) is an inclusion in the study. During this visit assess adherence to medication therapy General and to specific medications. The main factors affecting treatment adherence will be identified.

The second visit (V2) is planned for each patient 1 year after the first visit (V2). During the second visit the adherence to the therapy and frequency of Secondary Outcome Measures will be estimated. Impossible to visit repeated, a telephone interview can be done

ELIGIBILITY:
Inclusion Criteria:

* All patients with documented Сhronic heart failure who were included in register PROFILE from from Junuary 1, 2016 to July 31, 2020
* Ejection fraction <50% or
* Ejection fraction ≥ 50% plus increase of BNP>500 ng/l or NT-proBNP <50 years - 450 ng/l , 50-75 years > 900 ng/l; >75years > 1800 ng/l

Exclusion Criteria:

* Patients whose life status is defined as "dead"
* Patients who refused to participate in our study
* Refusal to sign informed agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with documented HF having consequentially come for consultation to the specialized cardiology department of the scientific research center from Junuary 1, 2016 to July 31, 2020 (Included in the registry PROFILE)
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Adherence to life-modifying treatment | 1 year
  The Adherence scale of the Russian National Society of evidence based pharmacotherapy will be used to assess patients' adherence to treatment. The patients will be asked questions about taking prescribed medications as recommended by a doctor.
  The score system with the min value in the scale 0 and the max value 4 is used for the assessment of the results: 0 - adherent, 1-2 - partially adherent, 3 - partially non-adherent, 4 - non adherent.

SECONDARY OUTCOMES:
Death | 1 year
  Total number - of all events
Chronic heart failure decompensation with hospitalization | 1 year
  Total number - of all events
Chronic heart failure decompensation without hospitalization | 1 year
  - onset of new symptoms (example:. Cardiac asthma, orthopnea- if you haven't registered before); -- increase in NYHA ≥1;- increase dose of diuretic
Myocardial Infarction | 1 year
  Total number - of all events
Unplanned hospitalization for Cardiovascular disease | 1 year
  Total number - of all events

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Martsevich, PhD, Study Chair — National Research Center for Preventive Medicine
Locations (1):
- Federal State Institution "National Medical Research Center for Preventive Medicine" of the Ministry of Healthcare of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martsevich SY, Lukina YV, Kutishenko NP, Guseynova ET. 0Effects of the COVID-19 Pandemic on Treatment Adherence in Patients with Chronic Heart Failure. Caspian J Intern Med. 2022;13(Suppl 3):199-203. doi: 10.22088/cjim.13.0.199. PMID 35872693